CLINICAL TRIAL: NCT06655363
Title: Anatomo-radiological Study of the Ankle's Lateral Ligament
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN762024/CHUSTE
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Ankle Injuries and Disorders
Keywords: Ankle; Subtalar instability; MRI; Anatomy
MeSH Terms: conditions — Ankle Injuries; Disease | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Anatomical arm
  Interventions: Other: Anatomical description
- Radiological arm
  Interventions: Other: Radiological (MRI) description

INTERVENTIONS:
Other: Anatomical description — Anatomical description of cervical ligament, calcaneo fibular ligament, interosseus talo-calcaneal ligament, talo-fibular ligament.
  Groups: Anatomical arm
Other: Radiological (MRI) description — Radiological (MRI) description of cervical ligament, calcaneo fibular ligament, interosseus talo-calcaneal ligament, talo-fibular ligament.
  Groups: Radiological arm

SUMMARY:
Subtalar instability is found in 30% of cases following a severe ankle sprain. Treatment is conditioned by subtalar involvement, so detection is essential. There is no consensus on the ligament anatomy of the subtalar region, making precise diagnosis of subtalar ligament damage difficult. The aim of this study is to provide a detailed description of the anatomy of the subtalar ligaments of interest, followed by a detailed radiological description (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with no history of sprain on studied ankle

Exclusion Criteria:

* Sprain on studied ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine follow-up MRI one year after ankle ligament surgery will be included.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2024-09-06 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-11 (Actual)

PRIMARY OUTCOMES:
Cervical ligament length | Day : 1
  Anatomical description of cervical ligament, by length (mm).

SECONDARY OUTCOMES:
Calcaneo fibular ligament length | Day : 1
  Anatomical description of calcaneo fibular ligament, by length (mm).
Cervical ligament width | Day : 1
  Anatomical description of cervical ligament, by width (mm).
Calcaneo fibular ligament width | Day : 1
  Anatomical description of calcaneo fibular ligament, by width (mm).
Calcaneo fibular ligament thickness | Day : 1
  Anatomical description of cervical calcaneo fibular ligament, by thickness (mm).
Cervical ligament thickness | Day : 1
  Anatomical description of cervical ligament, by thickness (mm).
Interosseus talo-calcaneal ligament length | Day : 1
  Anatomical description of interosseus talo-calcaneal ligament, by length (mm).
Interosseus talo-calcaneal ligament width | Day : 1
  Anatomical description of interosseus talo-calcaneal ligament, by width (mm).
Interosseus talo-calcaneal ligament thickness | Day : 1
  Anatomical description of interosseus talo-calcaneal ligament, by thickness (mm).
Talo-fibular ligament length | Day : 1
  Anatomical description of talo-fibular ligament, by length (mm).
Talo-fibular ligament width | Day : 1
  Anatomical description of talo-fibular ligament, by width (mm).
Talo-fibular ligament thickness | Day : 1
  Anatomical description of talo-fibular ligament, by thickness (mm).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Henri VERMOREL, MD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No